CLINICAL TRIAL: NCT00813657
Title: Effects of Resistance Exercise Training Program Performed During the 2nd and 3rd Trimesters of Pregnancy on Maternal and Newborn Health
Brief Title: Resistance Exercise Training During Pregnancy: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Ruben Barakat, Facultad de Ciencias de la Actividad Física y del Deporte - INEF, Universidad Politécnica de Madrid, Madrid, Spain
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 01562; 01562
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Gestational Age; Birth Weight; Anaemia; Gestational Diabetes Mellitus; Type of Delivery
MeSH Terms: conditions — Birth Weight; Anemia; Diabetes, Gestational | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Women in the intervention group were enrolled in three sessions/week of individually supervised, resistance exercise training performed over the second and third trimester of pregnancy (in total 26 weeks, ~80 training sessions). Heart rate (HR) was carefully and individually controlled (≤80% of age-predicted maximum HR value, 220-age) through a heart rate monitor during the training sessions. In brief, each session consisted of 35-40 minutes of exercise divided in a light intensity (≤60% maximal heart rate) warm-up period (~8 minutes), followed by toning and very light resistance exercises (~20 minutes) and a light intensity cool-down (~8 minutes) period. Resistance exercises were performed with barbells (≤3kg per exercise) or low-to-medium resistance bands (Therabands).

SUMMARY:
The investigators investigated the effects of a supervised maternal exercise training program (performed during the 2nd and 3rd trimesters of pregnancy) on maternal-newborn unit health outcomes in a group of previously sedentary healthy women. A matched control group was assessed over the same time period. Given the fact that most studies in the field have used aerobic exercises, here the investigators largely focused on very light resistance, toning exercises.

ELIGIBILITY:
Inclusion Criteria:

* sedentary (not exercising >20 minutes on >3 days per week)
* with singleton
* not at high risk for preterm delivery (no more than one previous preterm deliveries)
* women planning to give birth in the same obstetrics hospital department (Hospital Severo Ochoa, Madrid, Spain)

Exclusion Criteria:

* not being under medical follow-up throughout the entire pregnancy period were not included in the study
* women having serious medical condition that prevent them from exercising safely

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2000-01; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)